CLINICAL TRIAL: NCT06805669
Title: Integrating Early Palliative Care in Advanced SARcoma Patients for Enhanced QUALITY of Life: the SARQUALITY Study
Brief Title: This is a Randomized Study of Early Involvement of Palliative Care Along Side Standard Treatment Versus Standard Treatment Alone in Newly Diagnosed Patients With Advanced or Metastatic Soft Tissue Sarcoma (SARQUALITY)
Acronym: SARQUALITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SARC-004
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma
Keywords: Sarcoma; Palliative Care
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Referral to Palliative Care (Experimental)
  Interventions: Other: Early referral to palliative care
- Standard Treatment (Other)
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: Early referral to palliative care — Participant will be referred to palliative care at start of systemic treatment
  Arms: Early Referral to Palliative Care
Other: Standard Treatment — Participants will be referred to palliative care upon appearance of uncontrollable symptoms.
  Arms: Standard Treatment

SUMMARY:
The goal of this study is to learn whether early referral to palliative care improves quality of life for patients with advanced sarcoma.

Participants enrolled in this study will complete quality of life questionnaires before starting their treatment, and every 6 weeks for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent.
* Have histologically documented advanced sarcoma, either locally advanced not amenable to curative treatment, or metastatic.
* Age ≥ 18 years.
* Have not received any previous systemic treatment with palliative intent for advanced sarcoma.
* Performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Life expectancy > 6 months.
* Willing/able to complete questionnaires.

Exclusion Criteria:

* Clinical evidence of cognitive impairment that would preclude the ability to provide informed consent and complete questionnaires, at investigator´s discretion.
* Patient in need of urgent home support services or symptom management through a palliative care team.
* Patient is being actively followed by a palliative care physician.
* Active psychiatric disorder or drug abuse.
* Insufficient English literacy to complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To determine the difference of Health Related Quality of Life (HRQoL) for sarcoma patients who receive early palliative care versus not | From enrollment/baseline to 12 weeks
  HRQoL will be assessed using ESAS-r (Edmonton Symptom Assessment System - revised) and EORTC QLQ-C30 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire C-30).

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni R. Abdul Razak, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared.